CLINICAL TRIAL: NCT05815199
Title: Effectiveness and Impact of Counseling Enhanced Using Electronic Cigarettes for Harm Reduction in People With Serious Mental Illness
Brief Title: E-cigarettes for Harm Reduction Among Smokers With Serious Mental Illness
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23-00124
Record Dates: First submitted 2023-04-04; First posted 2023-04-18 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Cigarette Smoking
Keywords: E-cigarettes; Harm reduction; Cigarette smoking; Serious mental illness
MeSH Terms: conditions — Cigarette Smoking; Vaping; Harm Reduction | interventions — Electronic Nicotine Delivery Systems; Nicotine Replacement Therapy; elastin microfibril interface located protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- E-cigarettes (EC) (Experimental): Adult cigarette smokers with a SMI diagnosis randomized to the EC arm will receive NRT including nicotine patches and lozenges. Participants will also receive telehealth motivational counseling during the intervention period of 8 weeks.
  Interventions: Other: E-cigarette (EC); Behavioral: Harm-Reduction Counseling; Behavioral: Ecological Momentary Intervention (EMI) Text Messaging
- Nicotine Replacement Therapy (NRT) (Active Comparator): Adult cigarette smokers with a SMI diagnosis randomized to the NRT arm will receive NRT including nicotine patches and lozenges gum. Participants will also receive telehealth motivational counseling during the intervention period of 8 weeks.
  Interventions: Other: Nicotine Replacement Therapy (NRT); Behavioral: Harm-Reduction Counseling; Behavioral: Ecological Momentary Intervention (EMI) Text Messaging

INTERVENTIONS:
Other: E-cigarette (EC) — Fixed dose. Participants are to use the EC as replacement for smoking combustible cigarettes. Participants will vape the EC.
  Other Names: NJOY Ace or NJOY Daily Electronic Cigarette
  Arms: E-cigarettes (EC)
Other: Nicotine Replacement Therapy (NRT) — Includes nicotine patches and lozenges. NRT use recommendations will follow the guidelines of the product, e.g. one patch per day.
  Arms: Nicotine Replacement Therapy (NRT)
Behavioral: Harm-Reduction Counseling — At baseline, after randomization, participants will receive their first telehealth session (20~25 minutes) from a counselor trained in motivational interviewing, harm reduction, and smoking cessation. Up to five additional sessions will be delivered, 15~20 minutes each.
Behavioral: Ecological Momentary Intervention (EMI) Text Messaging — EMI can be defined as delivering tailored interventions via electronic messages (i.e., regular text messages) that include personalized feedback based on real-time assessment responses and other contextual factors. EMI will take place throughout the intervention period.

SUMMARY:
In this open-label, randomized controlled trial study, participants who smoke combustible cigarettes (CC) and are diagnosed with Serious Mental Illness (SMI) will be randomized in two arms to receive harm-reduction counseling and Ecological Momentary Intervention text messaging (EMI) along with either e-cigarettes (EC) or nicotine replacement therapy (NRT) such as patch and lozenges to compare the efficacy in CC smoking reduction.

ELIGIBILITY:
Inclusion Criteria:

* Currently smokes 5 or more CPD
* Willingness and ability to provide informed consent
* Age of at least 21 years
* Has SMI diagnosis (such as Schizophrenia, Schizoaffective disorders, Bipolar disorder, Depressive disorders, Trauma and stressor related disorders etc.) as determined using the MINI tool
* Interested in reducing CC smoking but not necessarily trying to quit
* Own a mobile phone or have regular access to a mobile phone
* Able to provide an additional contact to improve follow-up rates

Exclusion Criteria:

* Is pregnant or breastfeeding
* Used tobacco other than CC in the past 2 weeks (e.g., EC, cigarillo)
* Currently engaged in an attempt to quit CC
* Change in dose of their psychotropic medication(s) in the last 30 days
* Meeting DSM-V criteria for current alcohol or substance use disorder except for nicotine use disorder and active mild alcohol or substance use disorders.
* Past month suicidal ideation/suicide attempt and/or psychiatric hospitalization in the last 30 days

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-11-13 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants who Achieve a 100% Reduction in Cigarettes Per Day (CPD) by Week 4 | Up to Week 4
  Measured via self-report (daily diary about smoking behavior) and verified by exhaled carbon-monoxide (eCO) level (< 6 ppm).
Percentage of Participants who Achieve a 100% Reduction in Cigarettes Per Day (CPD) by Week 8 | Up to Week 8
  Measured via self-report (daily diary about smoking behavior) and verified by exhaled carbon-monoxide (eCO) level (< 6 ppm).

SECONDARY OUTCOMES:
Percentage of Participants who Achieve a 100% Reduction in Cigarettes Per Day (CPD) by Week 12 | Up to Week 12
  Measured via self-report (daily diary about smoking behavior) and verified by exhaled carbon-monoxide (eCO) level (< 6 ppm).
Self-Reported Percent Change in CPD from Baseline to Week 8 | Baseline, Week 8
  Measured via self-report (daily diary about smoking behavior).
Self-Reported Percent Change in CPD from Baseline to Week 12 | Baseline, Week 12
  Measured via self-report (daily diary about smoking behavior).
Change in American Thoracic Questionnaire Score from Baseline to Week 12 | Baseline, Week 12
  8-item questionnaire assessing general thoracic pain. Items are rated on a Likert scale from 1 (never) to 5 (every day). The total score is the sum of responses and ranges from 8-40; higher scores indicate more severe impact of general thoracic pain.
Change in Symptom Check Questionnaire Score from Baseline to Week 12 | Baseline, Week 12
  9-item assessment of chronic obstructive pulmonary disease (COPD) symptoms. Each item is marked as either "yes" or "no." The total score is the number of "yes" responses and ranges from 0-9; higher scores indicate more severe COPD symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Omar El-Shahawy, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request or for individual participant data meta-analysis beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data or researcher who provides a methodologically sound proposal executes a data use agreement with NYU Langone Health. Requests may be directed to: Omar.ElShahawy@nyulangone.org. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data or researchers who provide a methodologically sound proposal will be granted access upon reasonable request or for individual participant data meta-analysis. Requests should be directed to Omar.ElShahawy@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.